CLINICAL TRIAL: NCT03697928
Title: Searching for Non-invasive Magnetic Resonance-based Markers for CrAT Protein Activity and Carnitine Availability in Skeletal Muscle
Brief Title: Markers of Carnitine Acetyltransferase (CrAT) Protein Activity and Carnitine Availability
Status: Completed | Type: Observational
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Other Study IDs: NL63005.068.18
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Metabolism and Nutrition Disorder; Metabolic Disturbance
Keywords: Acetylcarnitine kinetic; Phosphocreatine (PCr) kinetic
MeSH Terms: conditions — Nutrition Disorders; Pathologic Complete Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — muscle biopsies
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CrAT subjects: 13 healthy adult men, with a wide range of maximal aerobic capacity will be included.
  Subjects will be classified as trained, physical active and untrained according to their VO2max.
  Subject will perform one-legged knee extension and flexion exercise inside the MRS scanner and cycling outside the scanner
  Interventions: Other: Exercise metabolism

INTERVENTIONS:
Other: Exercise metabolism — Participants will perform a series of exercises inside and outside the MRS/MRI scanner.

SUMMARY:
This study aims to measure skeletal muscle metabolism in vivo during exercise using the non-invasive Magnetic Resonance Spectroscopy (MRS) technique. Specifically, phosphocreatine (PCr) kinetic and Acetylcarnitine levels will be determined at resting, during exercise and during the recovery post exercise. The target population is adult healthy men, with a wide range of maximal physical capacity.

DETAILED DESCRIPTION:
Skeletal muscle mitochondrial activation during the transition from resting metabolism to exercise may modulated by CrAT activity. Furthermore, dynamic changes in acetylcarnitine during the transition from exercise to resting metabolism (acetylcarnitine off-kinetic) may also reflect the action of CrAT protein. To date, the only possibility to get information on CrAT activity is by taking a muscle biopsy and perform enzyme activity assays ex vivo. By dynamic MRS scanning, it might be possible to deduce information that reflects CrAT activity, thereby making the biopsy sampling unnecessary.

ELIGIBILITY:
Inclusion Criteria:

* Males, Generally healthy
* Age 18-40 years old
* BMI 18 - 25 kg/m2
* No medication use that interfere with the aims of the study
* Stable level of daily physical activity or training for at least 6 months

Exclusion Criteria:

* Females
* Regular smokers, drug abuse
* Participation in other studies
* Weight gain/loss > 3 kg in the last 6 months
* Contraindications for MRS scans:
* Vegetarian eating behavior

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In this study, 13 healthy young males (BMI <25 kg/m2), aged 18-40yr with different maximal aerobic capacity will be included. Specifically, 4 volunteers with a VO2max <40 ml/kg/min, 5 volunteers with a VO2max between 41 and 50 ml/kg/min and 4 volunteers with a VO2max >50 ml/kg/min will be included.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle PCr on-kinetic during exercise and carnitine acetyltransferase (CrAT) protein content/activity | MRS+Exercise test day 2
  The correlation between skeletal muscle PCr on-kinetic during one-legged exercise and CrAT protein activity will be determined.

SECONDARY OUTCOMES:
Skeletal muscle acetylcarnitine recovery after one-legged exercise and carnitine acetyltransferase (CrAT) protein content/activity | MRS+Exercise test day 2
  The correlation between skeletal muscle acetylcarnitine off-kinetic after one-legged exercise and CrAT protein activity will be determined.
Skeletal muscle CrAT protein activity, from muscle biopsy, and PCr breakdown rate during one-legged exercise | MRS+Exercise test day 1
  The correlation between CrAT protein activity and PCr hydrolysis/breakdown will be determined
Skeletal muscle acetylcarnitine formation capacity upon exercise and total carnitine availability in skeletal muscle | MRS+Exercise test day 2
  The correlation between acetylcarnitine formation upon exercise and total carnitine availability will be determined
Skeletal muscle mitochondrial function in vitro | MRS+Exercise test day 2
  The association between Skeletal muscle mitochondrial function in vitro and in vivo
Skeletal muscle oxygen availability | MRS test day 1
  in vivo assessment of oxygen availability in muscle tissue upon hypoxic stimulus during resting

CONTACTS AND LOCATIONS:
Overall Officials: Vera Schrauwen-Hinderling, Phd, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mancilla R, Pava-Mejia D, van Polanen N, de Wit V, Bergman M, Grevendonk L, Jorgensen J, Kornips E, Hoeks J, Hesselink MKC, Schrauwen-Hinderling VB. Invasive and noninvasive markers of human skeletal muscle mitochondrial function. Physiol Rep. 2023 Jun;11(12):e15734. doi: 10.14814/phy2.15734. PMID 37340318